CLINICAL TRIAL: NCT04251494
Title: An Observational, Cross-sectional Study Into the Future Cardiovascular Disease (CVD) Risk of Phenylketonuria (PKU) Patients on a Low Phenylalanine Treatment Diet (LPD).
Brief Title: A Study Into the Future Cardiovascular Disease (CVD) Risk of Phenylketonuria (PKU) Patients on a Low Phenylalanine Treatment Diet (LPD).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 254922
Record Dates: First submitted 2019-09-25; First posted 2020-02-05 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-01

CONDITIONS: Phenylketonurias; Cardiovascular Diseases
Keywords: PKU; CVD; Cardiovascular disease risk
MeSH Terms: conditions — Phenylketonurias; Cardiovascular Diseases | interventions — Ankle Brachial Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Routine blood samples from PKU participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phenylketonuria (PKU) participants: During their outpatient clinic appointment, participants will:
  * Undergo routine height and weight measurements and blood tests. A full patient history will be taken, including a record of cardiovascular disease within the family. Blood samples will be collected, including phenylalanine, lipids, vitamin B12 and related biomarkers.
  * Complete a 14-item diet history questionnaire, and fill in a 3 day diet diary before they arrive at their outpatient clinic appointment, which will be collected after the participant signs the informed written consent form.
  * Undergo assessment of carotid Intima-media thickness (CIMT), pulse wave velocity (PWV), ankle brachial pressure index (ABPI) and systolic and diastolic blood pressure.
  Interventions: Diagnostic Test: Carotid intima media thickness measurement (CIMT); Diagnostic Test: Pulse Wave Velocity measurement; Diagnostic Test: Ankle-brachial pressure index (ABPI); Other: Diet questionnaire and diet diary; Other: Routine blood samples
- Age and gender matched reference controls: Only Phenylketonuria (PKU) patients will be studied. Controls are generated from the literature. Reference CIMT values exist for a healthy population based on age and gender (Engelen et al., 2013), eliminating the need to assess age- and gender-matched controls. The study would otherwise require performing blood tests and vascular assessments on healthy individuals, generating a risk of harm and a possible incidental finding. It would be inconvenient for controls because they would need to travel to hospital and undergo invasive venepuncture.

INTERVENTIONS:
Diagnostic Test: Carotid intima media thickness measurement (CIMT) — CIMT is a measurement of the thickness of the two inner layers of the common carotid artery wall. Using ultrasound, a linear array transducer is placed on the surface of the skin at the neck. Electrocardiogram(ECG) electrodes are placed on each wrist and one on the ankle. An image of the common carotid artery (CCA) is then produced in anterior, posterior and lateral views, and saved along with the ECG recording. The wall thickness can then be measured at the same point in the cardiac cycle using semi-automated detection software (Philips QLAB), which can reduce observer variability. The CIMT will be averaged across left and right CIMTs, as the control reference values use an average of both sides.
  Groups: Phenylketonuria (PKU) participants
Diagnostic Test: Pulse Wave Velocity measurement — The PWV measures the speed of a pulse wave travelling between two points in the vascular systems of known distance between them. PWV will be measured by the gold standard carotid-femoral PWV method which is a direct measurement of aortic stiffness. A 3-Lead ECG is connected alongside measurements of the blood velocity trace for the left CCA 2cm proximal to the bifurcation, and for the left common femoral artery origin.
  Groups: Phenylketonuria (PKU) participants
Diagnostic Test: Ankle-brachial pressure index (ABPI) — A blood pressure cuff is placed around the ankle and upper arm of the participant. A continuous wave Doppler probe is used over the surface of the skin to locate the artery distal to the cuff (such as the brachial artery in the arm, or the anterior tibial and posterior tibial arteries in the ankle). The cuff is then inflated, and the systolic pressure identified by listening cessation of the sounds produced by the probe corresponding to blood flow in the artery. The ABPI is then the ratio of the highest systolic ankle pressure divided by the highest systolic brachial pressure for the left and right sides of the body.
  Groups: Phenylketonuria (PKU) participants
Other: Diet questionnaire and diet diary — Dietary information will be collected in two formats. One will be a 14-item questionnaire (Martínez-González et al., 2012), which is a simplified version of a comprehensive food frequency questionnaire. This provides a quick measure of compliance to a Mediterranean dietary pattern and a rough measure of protective and adverse dietary factors that could affect individual CVD risk. The second will be a 3-day diet diary (3DDD). This will consist of participants recording the foods that they consume and the quantities, which will then be analysed for macro- and micronutrient composition once completed.
  Groups: Phenylketonuria (PKU) participants
Other: Routine blood samples — Blood samples will be taken from participants during their outpatient appointment. Patients routinely have blood samples taken during this clinic. The study will use the results from the routine blood tests, and also extra blood samples to collect data on other biomarkers. The laboratory facilities at Guy's and St Thomas Hospitals will be used to conduct analysis, no other laboratories will be used. Data will be collected on Phenylalanine levels, lipids, vitamin B12 and related biomarkers.
  Groups: Phenylketonuria (PKU) participants

SUMMARY:
This study will assess the cardiovascular disease (CVD) risk in Phenylketonuria (PKU) patients on a low-phenylalanine diet (LPD).

Ultrasound tests, diet information and routine blood samples will be collected once per patient at their next outpatient appointment.

32 adults with PKU will be studied and compared to reference data for healthy people. The results will show if the PKU CVD risk differs from healthy people, and if CVD risk varies within people with PKU.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the largest cause of deaths worldwide each year. Many factors affect CVD including diet, genetics, exercise and smoking. It is unclear if Phenylketonuria (PKU) and the low-phenylalanine diet (LPD) affect CVD risk.

CVD risk can be predicted by measuring the thickness of the artery wall in the neck which supplies blood to the head. Thickness is measured using a non-invasive, safe ultrasound test (similar to pregnancy jelly scans). A wall thicker than normal indicates an increased CVD risk. A wall thinner than normal indicates a lower CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* Phenylketonuria patients at Guys and St Thomas' Centre for Inherited Metabolic Diseases, who have a diagnosis of Phenylketonuria at birth (following the introduction of the newborn screening programme), and who are over the age of 18 will be invited to take part in the study.
* The study will only include patients diagnosed at birth, which will allow a better assessment of the effects of the diet, which are not influenced by a late diagnosis and a prior diet which is not low-Phenylalanine.

Exclusion Criteria:

* Phenylketonuria patients at Guys and St Thomas' Centre for Inherited Metabolic Diseases, who have a diagnosis of Phenylketonuria after birth (not diagnosed during newborn screening), will be excluded from taking part in the study.
* If patients are pregnant, or plan to be pregnant during the study they will also be excluded.
* Patients with a previous history of cardiovascular disease, and/or a history of cardiovascular disease in their immediate family will also be excluded.
* Patients that are unable to understand and consent to the study (i.e. due to language issues or lacking capacity) will also be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Phenylketonuria patients at Guys and St Thomas' Centre for Inherited Metabolic Diseases, who have a diagnosis of Phenylketonuria at birth (following the introduction of the newborn screening programme), and who are over the age of 18 will be invited to take part in the study.
  The population is predominantly caucasian and middle aged.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2019-02-23 (Actual); Primary Completion 2021-04-22 (Estimated); Study Completion 2021-04-22 (Estimated)

PRIMARY OUTCOMES:
A single carotid-intima media thickness (CIMT) measurement in Phenylketonuria (PKU) participants and the corresponding age- and gender-matched controls. | 10 minutes
  A single CIMT measurement in PKU participants at their most recent outpatient appointment, and the corresponding age- and gender-matched CIMT, generated from the male (1) or female (2) equation for a healthy population using each participants' age and gender (Engelen et al., 2013).

SECONDARY OUTCOMES:
Pulse Wave Velocity (PWV) | 10 minutes
  will be compared to PKU patient biomarkers (median annual Phenylalanine levels, biomarkers and dietary factors) to assess if there is any correlation between compliance to diet and variation in cardiovascular risk within PKU patients.
Ankle brachial pressure index (ABPI) | 10 minutes
  will be compared to PKU patient biomarkers (median annual Phe levels, biomarkers and dietary factors) to assess if there is any correlation between compliance to diet and variation in cardiovascular risk within PKU patients.
Vitamin B12 levels from blood sample | 5 minutes
  will be compared to PKU patient measures (PWV, ABPI and CIMT) to assess if there is any correlation between compliance to diet and variation in cardiovascular risk within PKU patients.
Blood Phenylalanine levels | 5 minutes
  will be compared to PKU patient measures (PWV, ABPI and CIMT) to assess if there is any correlation between compliance to diet and variation in cardiovascular risk within PKU patients.
Blood low-density lipoprotein (LDL) cholesterol levels | 5 minutes
  will be compared to PKU patient measures (PWV, ABPI and CIMT) to assess if there is any correlation between compliance to diet and variation in cardiovascular risk within PKU patients.
Diet diary and diet questionnaire (Mediterranean Adherence Screener, 0-14 scale, 14 indicating full adherence, 0 indicating no adherence) | 3 days
  will be compared to PKU patient measures (PWV, ABPI and CIMT) to assess if there is any correlation between compliance to diet and variation in cardiovascular risk within PKU patients.

CONTACTS AND LOCATIONS:
Overall Officials: Radha Ramachandran, Principal Investigator — GSTT
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krikke M, Arends JE, Van Lelyveld S, Hoepelman A, Visseren F. Greater carotid intima media thickness at a younger age in HIV-infected patients compared with reference values for an uninfected cohort. HIV Med. 2017 Apr;18(4):275-283. doi: 10.1111/hiv.12428. Epub 2016 Aug 1. PMID 27477496
- [Background] Engelen L, Ferreira I, Stehouwer CD, Boutouyrie P, Laurent S; Reference Values for Arterial Measurements Collaboration. Reference intervals for common carotid intima-media thickness measured with echotracking: relation with risk factors. Eur Heart J. 2013 Aug;34(30):2368-80. doi: 10.1093/eurheartj/ehs380. Epub 2012 Nov 27. PMID 23186808
- [Background] Bots ML, Evans GW, Tegeler CH, Meijer R. Carotid Intima-media Thickness Measurements: Relations with Atherosclerosis, Risk of Cardiovascular Disease and Application in Randomized Controlled Trials. Chin Med J (Engl). 2016 Jan 20;129(2):215-26. doi: 10.4103/0366-6999.173500. PMID 26830994
- [Background] Hermida-Ameijeiras A, Crujeiras V, Roca I, Calvo C, Leis R, Couce ML. Arterial stiffness assessment in patients with phenylketonuria. Medicine (Baltimore). 2017 Dec;96(51):e9322. doi: 10.1097/MD.0000000000009322. PMID 29390507
- [Background] Htun P, Nee J, Ploeckinger U, Eder K, Geisler T, Gawaz M, Bocksch W, Fateh-Moghadam S. Fish-Free Diet in Patients with Phenylketonuria Is Not Associated with Early Atherosclerotic Changes and Enhanced Platelet Activation. PLoS One. 2015 Aug 20;10(8):e0135930. doi: 10.1371/journal.pone.0135930. eCollection 2015. PMID 26291823